CLINICAL TRIAL: NCT07389603
Title: Effect of a Restricted Time and Psychochrononutritional Feeding Intervention Program on the Nutritional Status of People With Metabolic Syndrome in Ciudad Guzmán.
Brief Title: Effects of Restricted-time and Psychochrononutritional Feeding in People With Metabolic Syndrome
Acronym: PSICRONUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Ana Patricia Zepeda Salvador, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP/T/36/25; DCAN/006/2025 (Other: Approval number of the Academic Board of the Doctorate in Behavioral Science with a focus on Food and Nutrition, Univer)
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Metabolic Syndrome
Keywords: Time restricted eating; Eating Behavior; Chrononutrition; Metabolic syndrome; Psychochrononutrition
MeSH Terms: conditions — Metabolic Syndrome; Intermittent Fasting; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal intervention group (Other): Participants will be instructed to adhere to a specific eating window, with flexibility to select their daily eating-window start and end times, as long as they fall within an 8- or 10-hour period. This intervention will last 8 weeks, during which they are instructed to consume all their caloric intake within the established time window.
  Interventions: Behavioral: Time restricted eating
- Grupo experimental (Experimental): Participants will be instructed to adhere to an 8- or 10-hour eating window, with flexibility to select their daily eating-window start and end times but must concentrate their caloric intake within that period. Additionally, the group receives a psychochrononutritional intervention consisting of weekly group sessions with an educational and behavioral focus for 8 weeks.
  Interventions: Behavioral: Time restricted eating; Behavioral: Psychochrononutritional intervention

INTERVENTIONS:
Behavioral: Time restricted eating — Behavioral and dietary intervention in which participants are instructed to consume all their food and caloric beverages within a fixed window (8 or 10 hours, depending on arm assignment). Outside of this window, only water or non-caloric beverages are permitted. The intervention will last 8 weeks.
  Other Names: Time restricted feeding
Behavioral: Psychochrononutritional intervention — Participants will receive a structured psychochrononutritional intervention consisting of eight weekly sessions. The program will cover the following topics:
  * Chrononutrition: The internal clock of eating.
  * Food groups and healthy menu planning.
  * Portion control: Learning to measure appropriately.
  * Effects of sugary drinks.
  * Sleep and its impact on eating habits.
  * Social and cultural factors in eating habits.
  * The relationship between physical activity and nutrition.
  * Making informed nutritional decisions.
  Arms: Grupo experimental

SUMMARY:
Metabolic syndrome is a cluster of risk factors, including abdominal obesity, high blood pressure, high triglycerides, and insulin resistance, that increase the risk of developing type 2 diabetes and cardiovascular disease. The prevalence of this syndrome is rising in Mexico. Recent research suggests that when we eat is as important as what we eat. Therefore, chrononutritional strategies such as time-restricted eating (TRE), where food intake is confined to a specific daily time window, have been developed and shown promising benefits. However, there are documented barriers to maintaining this nutritional strategy over time. Therefore, this study proposes that combining TRE with a psychochrononutritional program (integrating psychological, chronobiological, and nutritional components) will improve adherence to the nutritional strategy and lead to better health outcomes than only prescribing a specific eating window.

To this end, 64 adults (18-60 years old) with metabolic syndrome will be recruited in Ciudad Guzmán, Jalisco, Mexico. The TRE intervention will last eight weeks and include two groups. One group will undergo a psychochrononutritional intervention, whereas the other will receive only instructions regarding the eating window. Within each group, two subgroups will be formed: one assigned to an 8-hour eating window, and the other to a 10-hour window. Before and after the intervention, anthropometric, biochemical (lipid profile and plasma glucose), clinical (blood pressure), and dietary assessments will be performed. We expect reductions in blood pressure, glucose, triglycerides, and waist circumference as well as better adherence in the psychochrononutritional intervention group.

DETAILED DESCRIPTION:
Metabolic syndrome is a condition characterized by risk factors such as abdominal obesity, insulin resistance, hypertension, high triglycerides, and low HDL cholesterol. Together, these factors increase the likelihood of developing type 2 diabetes and cardiovascular disease. Given the growing prevalence of metabolic syndrome in Mexico and in the state of Jalisco, it is essential to develop strategies that contribute to its prevention and treatment.

Whitin this context, chrononutrition has gained prominence as evidence continues to show the benefits of aligning food intake with circadian rhythms. Time-Restricted Eating has been proposed as an effective strategy for preserving and maintaining the body's physiological health. Emerging evidence suggests it is an effective approach for individuals with metabolic syndrome, as it can improve glucose metabolism, reduce abdominal obesity, and lower the risk of developing metabolic syndrome.

The implementation of a restricted-time eating plan can be more effective when combined with a psychonutritional intervention, as this can improve adherence to the nutritional treatment and lead to better long-term results.

Therefore, this study aims to determine the effect of a restricted-time eating and a psychochrononutritional intervention program on the nutritional status of individuals with metabolic syndrome in Ciudad Guzmán, Jalisco. A randomized controlled trial will be conducted in adult residents, aged 18 to 60 years, of both sexes, diagnosed with metabolic syndrome. The sample size was calculated using a two-mean comparison equation, considering a 10% attrition rate. Resulting in a total sample of 64 participants, 32 for each group.

The study will be carried out in three phases. Phase one will include participants recruitment and confirmation of metabolic syndrome diagnosis. The second phase will integrate a baseline assessment, including anthropometric (weight, percentage of fat and muscle mass, waist circumference) and nutritional measurements, and questionnaires (diet quality index, the Chrononutrition Profile Questionnaire, adherence to treatment and the Pittsburgh Sleep Quality Index). The same variables will be evaluated at the end of the study. Participants will then complete an eight-week restricted-time eating intervention and will be assigned into two groups: one will receive psychonutritional support, and the other will only be given instructions regarding the eating window. Within each group, two subgroups will be created: one will have an 8-hour window, and the other a 10-hour eating window. The third phase will involve a follow up, measuring the same variables taken in phase one.

The data will be analyzed using the statistical software R. Descriptive analyses (means, standard deviations, frequencies, and percentages) will be calculated, followed by a normality test. A paired-samples t-test will be conducted to compare changes before and after the intervention in the following variables: a) anthropometric parameters: body weight, fat and muscle mass, and waist circumference; b) biochemical parameters: fasting plasma glucose, total cholesterol and fractions, and blood pressure; c) nutritional and behavioral variables: eating window and adherence to the eating schedule. In addition, an ANOVA or independent samples t-test will be performed to evaluate the differences between the groups: the group with psychochrononutritional intervention versus the group with minimal intervention, as well as the group with an 8-hour restricted eating window versus a 10-hour restricted eating window.

Expected outcomes include reductions in triglycerides, LDL cholesterol, fasting plasma glucose, blood pressure, and waist circumference, as well as an increase in HDL cholesterol. It is hypothesized that these improvements will be greater in the experimental groups, along with a higher adherence to the intervention. Collectively, these findings will help determine the effect of a time-restricted eating intervention combined with a psychochrononutritional approach and assess whether this strategy is a feasible option for improving metabolic health in patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 60 years
* Both sexes
* Feeding window ≥14 h/day
* Usual sleep duration >6.5 h
* Individuals diagnosed with metabolic syndrome who meet three or more of the criteria from Panel III of the National Cholesterol Education Program's Adult Treatment Guidelines:

  * Waist circumference: ≥102 cm for men, ≥88 cm for women
  * Triglycerides: ≥150 mg/dL or on treatment for hypertriglyceridemia
  * High-Density Lipoprotein (HDL) cholesterol: <40 mg/dL for men, <50 mg/dL for women
  * Blood pressure: systolic ≥130 mmHg and diastolic ≥85 mmHg or on treatment for hypertension
  * Fasting plasma glucose: ≥100 mg/dL
* Individuals who provide informed consent

Exclusion Criteria:

* (based on participant self-report unless medical records are available)

  * Pregnancy or lactation
  * Currently enrolled in a weight loss program
  * Current treatment with antidepressants, medications that affect glucose metabolism or appetite, or immunosuppressant therapy
  * History or presence of eating disorders
  * Sleep apnea

Elimination Criteria:

* Participants who do not attend more than two sessions of the psychochrononutritional intervention program.
* Participants who decide to withdraw their consent to continue in the study at any time for any reason.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Waist circumference | At the beginning (week 1) and end of the intervention (week 8).
  Measured in centimeters using a measuring tape at the level of the navel, at the end of a normal exhalation.
Blood Pressure | At the beginning (week 1) and end of the intervention (week 8).
  Measurement of systolic and diastolic blood pressure using a digital blood pressure monitor.
Glucose | At the beginning (week 1) and end of the intervention (week 8).
  Measurement of fasting plasma glucose, measured through a venous blood sample obtained between 7:30 and 8:30 am and processed using an automated colorimetric method.
HDL cholesterol | At the beginning (week 1) and end of the intervention (week 8).
  Measurement of HDL cholesterol measured through a venous blood sample obtained between 7:30 and 8:30 am and processed using an automated colorimetric method.
Triglycerides | At the beginning (week 1) and end of the intervention (week 8).
  Measurement of serum triglycerides measured through a venous blood sample obtained between 7:30 and 8:30 am and processed using an automated colorimetric method.
Treatment Adherence | Monitoring for 8 weeks.
  Degree to which participants follow the recommendations of the intervention program.

SECONDARY OUTCOMES:
Body weight | At the beginning (week 1) and end of the intervention (week 8).
  Measurement in kilograms using a digital scale. The participant should be barefoot, wearing as little clothing as possible, and preferably fasting.
Body composition analysis | At the beginning (week 1) and end of the intervention (week 8).
  Evaluation of fat and muscle mass relative to total body weight, expressed both as a percentage and in kilograms. This is determined using the bioelectrical impedance method.
Visceral fat | At the beginning (week 1) and end of the intervention (week 8).
  Adipose tissue located around the internal organs of the abdominal cavity. Measurement performed using bioelectrical impedance analysis.
Diet quality index | At the beginning (week 1) and end of the intervention (week 8).
  Assessment of overall nutritional quality based on dietary patterns. Score obtained using a dietary assessment tool (e.g., Healthy Eating Index).
Sleep quality | At the beginning (week 1) and end of the intervention (week 8).
  Subjective assessment of qualitative aspects such as sleep depth, daytime functioning, and recovery capacity, as well as identifying aspects such as duration, latency, and number of awakenings. Pittsburgh Sleep Quality Index questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yadira V Martínez Vázquez, PhD students, Study Chair — University of Guadalajara; Alma G Martínez Moreno, PhD, Study Chair — University of Guadalajara; César A Gómez Acosta, PhD, Study Chair — Universidad de Pamplona; Ana C Espinoza Gallardo, PhD, Study Chair — University of Guadalajara
Locations (1):
- Centro Universitario del Sur, Ciudad Guzmán, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No
For security and data protection reasons, access to participants' identities is restricted. Sharing identification forms with external researchers contradicts the principle of purpose limitation of consent, which stipulates that personal information will be treated anonymously and privately, ensuring that no data that could re-identify subjects is disclosed outside the authorized research team.

REFERENCES:
- [Background] Kozlov MM, Chernomordik LV. The protein coat in membrane fusion: lessons from fission. Traffic. 2002 Apr;3(4):256-67. doi: 10.1034/j.1600-0854.2002.030403.x. PMID 11929607